CLINICAL TRIAL: NCT03774875
Title: A Phase 4, Multi-center, Randomized, Double-blind, Placebo-controlled Study of the Impact of Apremilast (CC-10004) on Quality of Life, Efficacy, and Safety in Subjects With Manifestations of Plaque Psoriasis and Impaired Quality of Life
Brief Title: A Study of the Impact of Apremilast (CC-10004) on Quality of Life, Efficacy, and Safety in Adults With Manifestations of Plaque Psoriasis and Impaired Quality of Life
Acronym: EMBRACE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-10004-PSOR-020; U1111-1224-8381 (Registry Identifier: WHO); 2018-002850-58 (EudraCT Number)
Record Dates: First submitted 2018-12-11; First posted 2018-12-13 (Actual); Results first posted 2022-01-13 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Psoriasis
Keywords: Apremilast; CC-10004; Quality of life; Safety; Efficacy; Psoriasis manifestations
MeSH Terms: conditions — Psoriasis | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Apremilast 30 mg (Experimental): Participants will take apremilast 30 mg tablets orally twice a day for up to 52 weeks.
  Interventions: Drug: Apremilast
- Placebo / Apremilast 30 mg (Placebo Comparator): Participants will take placebo tablets orally twice a day for 16 weeks. After week 16, participants will be switched to receive apremilast 30 mg twice daily until Week 52.
  Interventions: Drug: Apremilast; Drug: Placebo

INTERVENTIONS:
Drug: Apremilast — Apremilast 30 mg tablets taken orally twice a day.
  Other Names: Otezla; CC-10004
Drug: Placebo — Placebo tablets taken orally twice a day
  Arms: Placebo / Apremilast 30 mg

SUMMARY:
The primary objective of the study is to assess the impact of treatment with apremilast 30 mg twice daily for 16 weeks, compared to placebo, on health-related quality of life (QOL) in adults with manifestations of plaque psoriasis and impaired quality of life.

DETAILED DESCRIPTION:
Participants will be randomized 2 (apremilast):1 (placebo) in approximately 10 countries in Western Europe. Participants will be block-randomized to each of the manifestations of psoriasis (scalp psoriasis, nail psoriasis, palmoplantar psoriasis, genital psoriasis, and psoriasis in visible locations). Participants presenting with multiple manifestations will be allocated to the manifestation which is most severe, as determined by the participant. All manifestations will be assessed for efficacy at each study visit.

The study will consist of 4 phases:

* Screening Phase - up to 5 weeks (35 days)
* Double-blind Placebo-controlled Phase - Weeks 0 to 16 Participants will receive treatment with either apremilast or matched placebo.
* Apremilast Extension Phase - Weeks 16 through 52 All participants will be switched to (or continue with) apremilast at week 16 and will maintain this dosing through week 52.
* Post-treatment Observational Follow-up Phase 4-week post-treatment observational follow-up phase for all participants who complete the study on treatment or discontinue from the study treatment early.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject is ≥ 18 years of age at the time of signing the informed consent form (ICF).
2. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
3. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
4. Subject has diagnosis of chronic plaque psoriasis for at least 6 months prior to baseline, that cannot be controlled by topical therapy.
5. Subject has a PASI score ranging from ≥ 3 to ≤ 10 at baseline.
6. Subject has a DLQI score > 10 at baseline.
7. Subject has presence of ≥ 1 clinical manifestations of plaque psoriasis, defined as at least one of the following:

   1. Moderate to severe scalp psoriasis, defined as Scalp Physician Global Assessment (ScPGA) ≥ 3
   2. Nail psoriasis, defined as onycholysis and onychodystrophy in at least 2 fingernails
   3. Moderate to severe genital plaque psoriasis, defined as modified static Physicians Global Assessment of Genitalia (sPGA-G) ≥ 3
   4. Moderate to severe palmoplantar psoriasis, defined as Palmoplantar Psoriasis Physicians Global Assessment (PPPGA) ≥ 3
   5. Moderate to severe plaque psoriasis in visible locations (dorsal hand, face, neck, and hairline) with static Physicians Global Assessment (sPGA) ≥ 3
8. Subject must be in general good health (except for psoriasis) as judged by the Investigator, based on medical history, physical examination, and clinical laboratories.

   (NOTE: The definition of good health means a subject does not have uncontrolled significant co-morbid conditions.)
9. Subject must have failed to respond to, or be contraindicated to, or intolerant to other systemic therapy, including, but not limited to, cyclosporine, methotrexate, acitretin, psoralen and ultraviolet-A-light (PUVA) fumaric acid esters or biologic therapies.
10. Subjects (in Italy only) must be non-responder to, contraindicated to, or intolerant to other systemic therapy (including cyclosporine, methotrexate, or PUVA) AND also be contraindicated to, or intolerant to biologics.
11. Females of childbearing potential (FCBP) must have a negative pregnancy test at Screening and Baseline. While on investigational product and for at least 28 days after taking the last dose of investigational product, FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options described below:

Option 1: Any one of the following highly effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy; OR Option 2: Male or female condom (latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]) PLUS one additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.

NOTE: Option 2 may not be acceptable as a highly effective contraception option in all countries per local guidelines/regulations.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subject has any condition, including other inflammatory diseases or dermatologic conditions, which confounds the ability to interpret data from the study, including other types of psoriasis (ie, erythrodermic, or guttate), other than plaque psoriasis or inverse psoriasis.
2. Subject has history of drug-induced psoriasis.
3. Subject has arthritis that requires systemic treatment.
4. Subject unable to avoid use of tanning booths for at least 4 weeks prior to baseline and during study.
5. Subject is currently enrolled in any other clinical trial involving an investigational product.
6. Other than psoriasis, subject has history of clinically significant or uncontrolled disease (as determined by the Investigator), including the presence of laboratory abnormalities, cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic disease, or other major disease, which places the subject at unacceptable risk if he/she were to participate in the study
7. Prior history of suicide attempt at any time in the subject's lifetime prior to signing the informed consent, or major psychiatric illness requiring hospitalization within the last 3 years prior to signing the informed consent.
8. Subjects with severe renal impairment, defined by estimated glomerular filtration rate (eGFR) or creatinine clearance (CLcr) less than 30 mL/min, are also categorized as having Stage 4 chronic kidney disease (CKD), and are excluded from the study.
9. Malignancy or history of malignancy or myeloproliferative or lymphoproliferative disease within the past 3 years, except for treated (ie, cured) basal cell or squamous cell in situ skin carcinomas.
10. Bacterial infections requiring treatment with oral or injectable antibiotics, or significant viral or fungal infections, within 4 weeks of Screening. Any treatment for such infections must have been completed and the infection cured, at least 4 weeks prior to Screening and no new or recurrent infections prior to the Baseline Visit.
11. Subject has received a live vaccine within 3 months of baseline or plans to do so during study.
12. Subject is a pregnant or breastfeeding (lactating) woman.
13. Subject has used topical therapy within 2 weeks of randomization (including, but not limited to, topical corticosteroids, retinoids or vitamin D analog preparations, tacrolimus, pimecrolimus, anthralin/dithranol, or moisturizers which contain urea or salicylic acid). Use of phototherapy within 4 weeks prior to randomization. Use of conventional systemic therapy or systemic corticosteroids within 4 weeks prior to randomization, except for conditions other than psoriasis or psoriatic arthritis. Use of biologic therapy within 5 pharmacokinetic half-lives.
14. Prior treatment with apremilast, or participation in a clinical study, involving apremilast.
15. Subject has any condition that confounds the ability to interpret data from the study.
16. Subject has history of allergy or hypersensitivity to any components of the IP (including placebo).
17. Subject has rare hereditary problem of galactose intolerance, lapp lactase deficiency or glucose-galactose malabsorption.
18. Subject's most severe manifestation corresponds to a manifestation whose randomization block has already been fully enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (67):
- France (10):
  - Research Site, Bordeaux
  - Research Site, Grenoble
  - Research Site, Lyon
  - Research Site, Paris
  - Research Site, Pringy
  - Research Site, Rouen
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Toulouse
  - Research Site, Valence
  - Research Site, Valenciennes
- Germany (18):
  - Research Site, Aachen
  - Research Site, Augsburg
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Bonn
  - Research Site, Erlangen
  - Research Site, Frankfurt am Main
  - Research Site, Gera
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Jena
  - Research Site, Kiel
  - Research Site, Langenau
  - Research Site, Lübeck
  - Research Site, Marburg
  - Research Site, München
  - Research Site, Tübingen
  - Research Site, Ulm
- Italy (8):
  - Research Site, Bologna
  - Research Site, Catania
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Napoli, Campania
  - Research Site, Perugia
  - Research Site, Roma
- Spain (12):
  - Research Site, Badalona, Catalonia
  - Research Site, Alcorcón, Madrid
  - Research Site, Fuenlabrada, Madrid
  - Research Site, Alicante, Valencia
  - Research Site, Manises, Valencia
  - Research Site, Castellon
  - Research Site, Lugo
  - Research Site, Madrid
  - Research Site, Murcia
  - Research Site, Salamanca
  - Research Site, Santiago de Compostela
  - Research Site, Seville
- Switzerland (2):
  - Research Site, Lausanne
  - Research Site, Zurich
- United Kingdom (17):
  - Research Site, Barnet
  - Research Site, Birmingham
  - Research Site, Brighton
  - Research Site, Bury St Edmunds
  - Research Site, Dumfries
  - Research Site, Dundee
  - Research Site, Exeter
  - Research Site, Gloucester
  - Research Site, Isleworth
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Newport
  - Research Site, Nottingham
  - Research Site, Plymouth
  - Research Site, Redhill
  - Research Site, Southampton
  - Research Site, Stourbridge

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Mrowietz U, Barker J, Conrad C, Jullien D, Gisondi P, Flower A, Reddy J, Paris M, Picard H, Jardon S, Augustin M. Efficacy and safety of apremilast in patients with limited skin involvement, plaque psoriasis in special areas and impaired quality of life: Results from the EMBRACE randomized trial. J Eur Acad Dermatol Venereol. 2023 Feb;37(2):348-355. doi: 10.1111/jdv.18689. Epub 2022 Nov 14. PMID 36300769
- [Background] Augustin M, Barker J, Conrad C, Jullien D, Carrascosa JM, Reddy J, Amouzadeh H, Colgan S, Zou H, Mrowietz U. Efficacy and Safety of Apremilast Over 52 Weeks in Patients with Plaque Psoriasis in High-Impact Areas and Impaired Quality of Life. Dermatol Ther (Heidelb). 2025 Jul;15(7):1915-1929. doi: 10.1007/s13555-025-01389-z. Epub 2025 May 3. PMID 40317400
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were enrolled at 55 centers in France, Germany, Italy, Spain, Switzerland, and the United Kingdom.
  The study consisted of a 16-week placebo-controlled period and a 36-week apremilast extension period.
Pre-assignment Details: Participants were randomized in a 1:2 ratio to receive placebo or apremilast. Participants were block-randomized to each of the manifestations of psoriasis (scalp psoriasis, nail psoriasis, palmoplantar psoriasis, genital psoriasis, and psoriasis in visible locations).
Groups:
- Placebo / Apremilast 30 mg: Participants received placebo tablets orally twice a day for 16 weeks. At Week 16 participants switched to receive 30 mg apremilast orally twice a day up to week 52.
- Apremilast 30 mg: Participants received apremilast 30 mg tablets orally twice a day for 52 weeks.
Period: Placebo-controlled Period (Week 1-16)
Arm/Group | Placebo / Apremilast 30 mg | Apremilast 30 mg
Started | 92 | 185
Received Study Drug | 91 | 185
Completed | 69 | 152
Not Completed | 23 | 33
Not completed — Adverse Event | 8 | 16
Not completed — Lack of Efficacy | 2 | 4
Not completed — Withdrawal by Subject | 12 | 10
Not completed — Lost to Follow-up | 0 | 2
Not completed — Protocol Deviation | 0 | 1
Not completed — Reason Unknown | 1 | 0
Period: Apremilast Extension Period (Week 16-52)
Arm/Group | Placebo / Apremilast 30 mg | Apremilast 30 mg
Started | 69 | 152
Completed | 53 | 105
Not Completed | 16 | 47
Not completed — Adverse Event | 6 | 9
Not completed — Lack of Efficacy | 2 | 11
Not completed — Withdrawal by Subject | 7 | 20
Not completed — Non-compliance with Study Drug | 0 | 2
Not completed — Other | 1 | 1
Not completed — Protocol Deviation | 0 | 1
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo / Apremilast 30 mg | Apremilast 30 mg | Total
Number analyzed (Participants) | 92 | 185 | 277
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (13.68) | 47.4 (14.28) | 48.6 (14.16)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 73 | 158 | 231
  ≥ 65 years | 19 | 27 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 79 | 114
  Male | 57 | 106 | 163
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 89 | 179 | 268
  Black or African American | 0 | 2 | 2
  Asian | 1 | 1 | 2
  Not Collected or Unknown | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  France | 6 | 13 | 19
  Germany | 45 | 102 | 147
  Italy | 8 | 11 | 19
  Spain | 23 | 24 | 47
  Switzerland | 1 | 7 | 8
  United Kingdom | 9 | 28 | 37
Duration of Plaque Psoriasis [Mean (Standard Deviation); unit: years] | 18.41 (13.350) | 16.31 (13.116) | 17.01 (13.207)
Primary Manifestations for Stratifications [Count of Participants; unit: Participants]
  Scalp Psoriasis | 23 | 45 | 68
  Nail Psoriasis | 20 | 40 | 60
  Palmoplantar Psoriasis | 10 | 22 | 32
  Genital Psoriasis | 15 | 28 | 43
  Psoriasis in Visible Locations | 24 | 50 | 74
Dermatology Life Quality Index (DLQI) Score [Mean (Standard Deviation); unit: score on a scale] — The DLQI is a 10-item skin disease-specific questionnaire used to evaluate the impact of skin disease on health-related quality of life (QOL). The items address symptoms and feelings, daily activities, leisure, work/school, personal relationships, and issues with treatment. Questions are answered on a 4-point scale from 0 (not at all/not applicable) to 3 (very much). Item scores are added to provide a total score from 0 to 30, with higher scores indicating greater impairment of QOL.
  score on a scale | 18.5 (4.94) | 18.1 (4.86) | 18.2 (4.88)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved a ≥ 4-point Reduction From Baseline in Dermatology Life Quality Index (DLQI) at Week 16
Description: The DLQI is a 10-item skin disease-specific questionnaire used to evaluate the impact of skin disease on health-related quality of life (QOL). The items address symptoms and feelings, daily activities, leisure, work/school, personal relationships, and issues with treatment. Questions are answered on a 4-point scale from 0 (not at all/not applicable) to 3 (very much). Item scores are added to provide a total score from 0 to 30, with higher scores indicating greater impairment of QOL.
Time Frame: Baseline and week 16
Population: All randomized participants; Missing data at week 16 were imputed using multiple imputation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo: Participants received placebo tablets orally twice a day for 16 weeks.
- Apremilast 30 mg: Participants received apremilast 30 mg tablets orally twice a day for 16 weeks.
Arm/Group | Placebo | Apremilast 30 mg
Number analyzed (Participants) | 92 | 185
percentage of participants | 41.3 [30.0 to 52.6] | 73.3 [66.7 to 79.9]
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; The CMH (Cochran-Mantel-Haenszel) test adjusting for the stratification of the 5 difficult to treat manifestation types at randomization; Adjusted Difference in Response Rates = 31.9, 95% CI 2-sided [18.6 to 45.2], Standard Error of Mean 6.78 — Adjusted difference (apremilast - placebo) in response rates calculated using the weighted average of the treatment differences across the strata with the CMH weights

2. Secondary Outcome: Change From Baseline in DLQI at Week 16
Description: The DLQI is a 10-item skin disease-specific questionnaire used to evaluate the impact of skin disease on health-related quality of life. The items address symptoms and feelings, daily activities, leisure, work/school, personal relationships, and issues with treatment. Questions are answered on a 4-point scale from 0 (not at all/not applicable) to 3 (very much). Item scores are added to provide a total score from 0 to 30, with higher scores indicating greater impairment of QOL. A negative change from baseline indicates improvement in quality of life.
Time Frame: Baseline and week 16
Population: All randomized participants; Missing data at week 16 were imputed using multiple imputation.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Apremilast 30 mg
Number analyzed (Participants) | 92 | 185
score on a scale | -3.4 (0.80) | -8.7 (0.54)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p < 0.0001, ANCOVA; ANCOVA model with treatment arm and stratification factor as independent variables and baseline value as a covariate; Least Squares (LS) Mean Difference = -5.3, 95% CI 2-sided [-7.15 to -3.43], Standard Error of Mean 0.95 — Difference in LS Means = Apremilast - Placebo

3. Secondary Outcome: Percent Change From Baseline in Body Surface Area (BSA) Affected by Psoriasis at Week 16
Description: Body surface area is a measurement of involved skin. The overall BSA affected by psoriasis was estimated based on the palm area of the participant's hand (entire palmar surface or "handprint"), which equates to approximately 1% of total BSA.
Time Frame: Baseline and week 16
Population: All randomized participants; Missing data at week 16 were imputed using multiple imputation.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Apremilast 30 mg
Number analyzed (Participants) | 92 | 185
percent change | 18.5 (12.95) | -19.8 (6.58)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.0085, ANCOVA; ANCOVA model with treatment arm and stratification factor as independent variables and the baseline value as a covariate variable; LS Mean Difference = -38.4, 95% CI 2-sided [-66.58 to -10.14], Standard Error of Mean 14.12 — LS Mean Difference = Apremilast - Placebo

4. Secondary Outcome: Change From Baseline in Itch Numeric Rating Scale (NRS) Score at Week 16
Description: The Itch Numeric Rating Scale (NRS) asked participants to assess the worst severity of itch experienced over the past 24 hours on an 11-point scale anchored from 0, representing 'no itching' to 10, representing 'worst itch imaginable'.
  A negative change from baseline indicates improvement in itch severity.
Time Frame: Baseline and week 16
Population: All randomized participants; Missing data at week 16 were imputed using multiple imputation.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Apremilast 30 mg
Number analyzed (Participants) | 92 | 185
score on a scale | -0.9 (0.32) | -2.5 (0.21)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p < 0.0001, ANCOVA; ANCOVA model with treatment arm and stratification factor as independent variables and the baseline value as a covariate; LS Mean Difference = -1.6, 95% CI 2-sided [-2.34 to -0.86], Standard Error of Mean 0.38 — LS Mean Difference = Apremilast - Placebo

5. Secondary Outcome: Change From Baseline in Skin Discomfort/Pain Visual Analog Scale (VAS) at Week 16
Description: Participants were asked to indicate their level of skin discomfort/pain in the past week by placing a vertical stroke on a 100 mm horizontal line on which the left-hand boundary (0) represents no skin discomfort/pain, and the right-hand boundary (100) represents worst possible skin discomfort/pain. The distance from the mark to the left-hand boundary was recorded.
  A negative change from baseline indicates improvement in skin discomfort/pain.
Time Frame: Baseline and week 16
Population: All randomized participants; Missing data at week 16 were imputed using multiple imputation.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Apremilast 30 mg
Number analyzed (Participants) | 92 | 185
score on a scale | -5.4 (3.61) | -21.5 (2.36)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.0003, ANCOVA; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -16.1, 95% CI 2-sided [-24.63 to -7.60], Standard Error of Mean 4.31 — LS Mean Difference = Apremilast - Placebo

6. Secondary Outcome: Percentage of Participants Who Achieved a Psoriasis Area Severity Index (PASI) Score < 3 at Week 16
Description: The PASI score is a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness, and scaling) and degree of skin surface area involvement on defined anatomical regions. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The total qualitative score (sum of erythema, thickness, and scaling scores) is multiplied by the degree of involvement for each anatomic region and then multiplied by a constant and the values for each anatomic region are summed to yield the PASI score. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity.
Time Frame: Week 16
Population: All randomized participants; missing data at week 16 were imputed using multiple imputation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Apremilast 30 mg
Number analyzed (Participants) | 92 | 185
percentage of participants | 26.3 [16.6 to 36.0] | 39.7 [32.3 to 47.1]
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.0328, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for the stratification of the 5 difficult to treat manifestation types at randomization; Adjusted Difference in Response Rates = 13.5, 95% CI 2-sided [1.1 to 25.8], Standard Error of Mean 6.30 — The adjusted difference in response rates (Apremilast - Placebo) using the weighted average of the treatment differences across the strata with the CMH weights

7. Secondary Outcome: Percentage of Participants Who Achieved a Patient Benefit Index (PBI) Global Score of ≥ 1 at Week 16
Description: The PBI is a validated patient-reported instrument to assess patient-relevant benefits of psoriasis treatment. Prior to starting study treatment, participants were asked to assess the importance of a series of treatment goals (from not important to very important) by completing the Patient Needs Questionnaire (PNQ). After a period of treatment (16 weeks), participants were then asked to assess the extent to which these goals were achieved (from not at all to very) by completing the Patient Benefit Questionnaire (PBQ). The Patient Benefit Index represents the benefits realized as a function of most important needs. The PBI score ranges from 0 (no benefit) to 4 (maximum benefit).
Time Frame: Week 16
Population: All randomized participants; Missing data at week 16 were imputed using multiple imputation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Apremilast 30 mg
Number analyzed (Participants) | 92 | 185
percentage of participants | 39.9 [28.8 to 51.0] | 76.6 [70.2 to 83.1]
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusting for the stratification of the 5 difficult to treat manifestation types at randomization; Adjusted Difference in Response Rates = 37.0, 95% CI 2-sided [24.1 to 49.9], Standard Error of Mean 6.58 — Adjusted difference (Apremilast - Placebo) in response rates using the weighted average of the treatment differences across the strata with the CMH weights

8. Secondary Outcome: Percent Change From Baseline in European Quality of Life 5-Dimension (EQ-5D) VAS Score at Week 16
Description: EQ-5D measures the participant's general health state on a vertical VAS and five quality of life domains. The EQ-5D VAS score ranges from 0 to 100, where a score of 0 indicates the worst imaginable health states and a score of 100 indicates the best imaginable health state. A positive change from baseline indicates improvement.
Time Frame: Baseline and week 16
Population: All randomized participants with available data at baseline and week 16.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Apremilast 30 mg
Number analyzed (Participants) | 70 | 160
percent change | 18.9 (15.96) | 33.8 (10.67)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.4216, ANCOVA; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = 14.9, 95% CI 2-sided [-21.62 to 51.48], Standard Error of Mean 18.55 — LS Mean Difference = Apremilast - Placebo

9. Secondary Outcome: Percent Change From Baseline in EQ-5D Index Score at Week 16
Description: EQ-5D measures the participants general health state as a vertical VAS and 5 quality of life domains: mobility, self-care, main activity (work, study, housework, family/leisure activities), pain/discomfort, and anxiety/depression. Each dimension is rated on three levels (no problems, some/moderate problems, extreme problems). An EQ-5D summary index is derived by applying a formula that attaches values (weights) to each of the levels in each dimension.
  EQ-5D index values were derived using the UK scoring algorithm, where a higher score indicates a better health state. The range of the score is from -0.224 to 1, with 0 corresponding to death, 1 corresponding to full health, and negative numbers indicate health states worse than death. A positive change from baseline indicates improvement.
Time Frame: Baseline and week 16
Population: All randomized participants with available data at baseline and week 16.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Apremilast 30 mg
Number analyzed (Participants) | 70 | 160
percent change | 165.9 (89.80) | 17.8 (59.59)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.1559, ANCOVA; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -148.024, 95% CI 2-sided [-352.8793 to 56.8304], Standard Error of Mean 103.9525 — LS Mean Difference = Apremilast - Placebo

10. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment Questionnaire: Psoriasis (WPAI: PSO) at Week 16: Percentage Work Time Missed
Description: The WPAI: PSO is a self-administered questionnaire designed to address impairment to the work productivity and activity of participants due to psoriasis in the past 7 days. Percent of work time missed is derived from the number of hours of work missed due to psoriasis symptoms as a percentage of total hours that should have been worked. A higher percentage indicates more hours missed, and a negative change from baseline indicates improvement.
Time Frame: Baseline and week 16
Population: All randomized participants with available data and who had reported being employed at baseline and at week 16.
Measure: Least Squares Mean (Standard Error); unit: percent impairment
Arm/Group | Placebo | Apremilast 30 mg
Number analyzed (Participants) | 36 | 104
percent impairment | -4.1 (2.56) | -0.9 (1.54)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.2667, ANCOVA; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = 3.1, 95% CI 2-sided [-2.43 to 8.73], Standard Error of Mean 2.82 — LS Mean Difference = Apremilast - Placebo

11. Secondary Outcome: Change From Baseline in WPAI: PSO at Week 16: Percentage Work Impairment
Description: The WPAI: PSO is a self-administered questionnaire designed to address impairment to the work productivity and activity of participants due to psoriasis in the past 7 days. Percent impairment while working was derived from the participant's assessment of the degree to which psoriasis affected their productivity while working. A higher percentage indicates greater impairment and less productivity, and a negative change from baseline indicates improvement.
Time Frame: Baseline and week 16
Population: All randomized participants with available data and who had reported being employed at baseline and at week 16.
Measure: Least Squares Mean (Standard Error); unit: percent impairment
Arm/Group | Placebo | Apremilast 30 mg
Number analyzed (Participants) | 36 | 102
percent impairment | -11.5 (3.82) | -13.9 (2.32)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.5620, ANCOVA; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -2.5, 95% CI 2-sided [-10.83 to 5.91], Standard Error of Mean 4.23 — LS Mean Difference = Apremilast - Placebo

12. Secondary Outcome: Change From Baseline in WPAI: PSO at Week 16: Percentage Overall Work Impairment
Description: The WPAI: PSO is a self-administered questionnaire designed to address impairment to the work productivity and activity of participants due to psoriasis in the past 7 days. Percent overall work impairment takes into account both hours missed due to psoriasis symptoms and the participant's assessment of the degree to which psoriasis affected their productivity while working. A higher percentage indicates greater impairment and less productivity, and a negative change from baseline indicates improvement.
Time Frame: Baseline and week 16
Population: All randomized participants with available data and who had reported being employed at baseline and at week 16.
Measure: Least Squares Mean (Standard Error); unit: percent impairment
Arm/Group | Placebo | Apremilast 30 mg
Number analyzed (Participants) | 36 | 104
percent impairment | -13.2 (4.35) | -13.8 (2.63)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.8927, ANCOVA; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.6, 95% CI 2-sided [-10.16 to 8.86], Standard Error of Mean 4.81 — LS Mean Difference = Apremilast - Placebo

13. Secondary Outcome: Change From Baseline in WPAI: PSO at Week 16: Percentage Activity Impairment
Description: The WPAI: PSO is a self-administered questionnaire designed to address impairment to the work productivity and activity of participants due to psoriasis in the past 7 days. Percent activity impairment is derived from the patient's assessment of the degree to which psoriasis affected their regular daily unpaid activities, measured on a VAS from 1 (no effect on daily activities) to 10 (psoriasis completely prevented daily activities). A higher percentage indicates greater impairment and less productivity, and a negative change from baseline indicates improvement.
Time Frame: Baseline and week 16
Population: All randomized participants with available data at baseline and at week 16.
Measure: Least Squares Mean (Standard Error); unit: percent impairment
Arm/Group | Placebo | Apremilast 30 mg
Number analyzed (Participants) | 42 | 116
percent impairment | -13.4 (3.66) | -21.2 (2.24)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.0572, ANCOVA; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -7.8, 95% CI 2-sided [-15.90 to 0.24], Standard Error of Mean 4.09 — LS Mean Difference = Apremilast - Placebo

14. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) During the Placebo-controlled Period
Description: An adverse event (AE) is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values, regardless of etiology. Any worsening of a preexisting condition was considered an AE.
  A serious adverse event (SAE) is any AE occurring at any dose that:
  * Resulted in death;
  * Was life-threatening;
  * Required inpatient hospitalization or prolongation of existing hospitalization;
  * Resulted in persistent or significant disability/incapacity;
  * Was a congenital anomaly/birth defect;
  * Constituted an important medical event. The Investigator assessed the severity/intensity of each event as mild, moderate, or severe based on level of symptoms.
Time Frame: From first dose of study drug to week 16 or up to 28 days after last dose for participants who didn't enter the apremilast extension period.
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Apremilast 30 mg
Number analyzed (Participants) | 91 | 185
Participants
  Any TEAE | 54 | 152
  Drug-related TEAE | 26 | 113
  Severe TEAEs | 1 | 10
  Serious TEAEs | 0 | 8
  Serious drug-related TEAE | 0 | 1
  TEAE leading to drug interruption | 0 | 9
  TEAE leading to drug withdrawal | 8 | 18
  TEAE leading to death | 0 | 0

15. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities During the Placebo-controlled Period
Description: Marked laboratory abnormalities are defined for each parameter below.
  ULN = upper limit of normal
Time Frame: 16 weeks
Population: All randomized participants who received at least one dose of study drug with at least one post-baseline measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Apremilast 30 mg
Number analyzed (Participants) | 80 | 162
Participants
  Alanine Aminotransferase > 3 × ULN: number analyzed (Participants) | 80 | 161
  Alanine Aminotransferase > 3 × ULN | 0 | 2
  Albumin < 25 g/L | 0 | 0
  Alkaline Phosphatase > 400 U/L | 0 | 0
  Aspartate Aminotransferase > 3 × ULN: number analyzed (Participants) | 79 | 160
  Aspartate Aminotransferase > 3 × ULN | 0 | 1
  Bilirubin (umol/L) > 1.8 × ULN: number analyzed (Participants) | 80 | 161
  Bilirubin (umol/L) > 1.8 × ULN | 0 | 0
  Blood Urea Nitrogen > 15 mmol/L | 0 | 2
  Calcium < 1.8 mmol/L | 0 | 0
  Calcium > 3.0 mmol/L | 0 | 0
  Cholesterol > 7.8 mmol/L | 0 | 1
  Creatinine > 1.7 × ULN | 0 | 1
  Glucose < 2.8 mmol/L | 0 | 0
  Glucose > 13.9 mmol/L | 0 | 3
  Hemoglobin A1C (Fasting) > 9%: number analyzed (Participants) | 35 | 97
  Hemoglobin A1C (Fasting) > 9% | 0 | 3
  Lactate Dehydrogenase > 3 × ULN: number analyzed (Participants) | 69 | 155
  Lactate Dehydrogenase > 3 × ULN | 0 | 0
  Potassium < 3.0 mmol/L: number analyzed (Participants) | 80 | 161
  Potassium < 3.0 mmol/L | 0 | 0
  Potassium > 5.5 mmol/L: number analyzed (Participants) | 80 | 161
  Potassium > 5.5 mmol/L | 0 | 1
  Sodium < 130 mmol/L: number analyzed (Participants) | 80 | 161
  Sodium < 130 mmol/L | 0 | 0
  Sodium > 150 mmol/L: number analyzed (Participants) | 80 | 161
  Sodium > 150 mmol/L | 0 | 0
  Triglycerides > 3.4 mmol/L | 6 | 6
  Hemoglobin: Female < 85 g/L, Male < 105 g/L: number analyzed (Participants) | 79 | 160
  Hemoglobin: Female < 85 g/L, Male < 105 g/L | 0 | 0
  Hemoglobin: Female > 170 g/L, Male > 185 g/L: number analyzed (Participants) | 79 | 160
  Hemoglobin: Female > 170 g/L, Male > 185 g/L | 0 | 0
  Leukocytes < 1.5 × 10^9/L: number analyzed (Participants) | 79 | 160
  Leukocytes < 1.5 × 10^9/L | 0 | 0
  Lymphocytes < 0.8 × 10^9/L: number analyzed (Participants) | 79 | 159
  Lymphocytes < 0.8 × 10^9/L | 1 | 2
  Neutrophils, Segmented < 1.0 × 10^9/L: number analyzed (Participants) | 79 | 159
  Neutrophils, Segmented < 1.0 × 10^9/L | 0 | 0
  Platelets < 75 × 10^9/L: number analyzed (Participants) | 79 | 159
  Platelets < 75 × 10^9/L | 0 | 1
  Platelets > 600 × 10^9/L: number analyzed (Participants) | 79 | 159
  Platelets > 600 × 10^9/L | 0 | 0

16. Secondary Outcome: Change From Baseline in Blood Pressure During the Placebo-controlled Period
Time Frame: Baseline, week 2, week 4, and week 16
Population: Randomized participants who received at least one dose of study drug and with a baseline value and a post-baseline value at each time point.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Apremilast 30 mg
Number analyzed (Participants) | 91 | 185
mmHg
  Systolic: week 2: number analyzed (Participants) | 88 | 174
  Systolic: week 2 | -0.5 (11.17) | 0.1 (12.44)
  Systolic: week 4: number analyzed (Participants) | 79 | 170
  Systolic: week 4 | 1.9 (12.29) | 0.4 (11.88)
  Systolic: week 16: number analyzed (Participants) | 67 | 153
  Systolic: week 16 | 2.2 (13.77) | 1.0 (12.66)
  Diastolic: week 2: number analyzed (Participants) | 88 | 174
  Diastolic: week 2 | -0.1 (7.89) | -0.6 (8.27)
  Diastolic: week 4: number analyzed (Participants) | 79 | 170
  Diastolic: week 4 | 1.3 (7.62) | -1.0 (9.51)
  Diastolic: week 16: number analyzed (Participants) | 67 | 153
  Diastolic: week 16 | 0.8 (8.29) | 0.6 (9.12)

17. Secondary Outcome: Change From Baseline in Pulse Rate During the Placebo-controlled Period
Time Frame: Baseline and week 2, week 4, and week 16
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Placebo | Apremilast 30 mg
Number analyzed (Participants) | 91 | 185
beats/minute
  Week 2: number analyzed (Participants) | 87 | 173
  Week 2 | 0.3 (10.82) | 3.4 (9.75)
  Week 4: number analyzed (Participants) | 79 | 170
  Week 4 | -0.4 (10.17) | 3.5 (10.43)
  Week 16: number analyzed (Participants) | 67 | 149
  Week 16 | 1.0 (9.97) | 2.0 (10.99)

18. Secondary Outcome: Change From Baseline in Body Weight During the Placebo-controlled Period
Time Frame: Baseline and week 2, week 4, and week 16
Population: Randomized participants who received at least one dose of study drug and with with a baseline value and a post-baseline value at each time point.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo | Apremilast 30 mg
Number analyzed (Participants) | 91 | 185
kg
  Week 2: number analyzed (Participants) | 88 | 174
  Week 2 | -0.02 (1.161) | -0.31 (1.188)
  Week 4: number analyzed (Participants) | 79 | 170
  Week 4 | 0.04 (1.285) | -0.57 (2.060)
  Week 16: number analyzed (Participants) | 67 | 153
  Week 16 | 0.08 (2.337) | -0.98 (2.722)

19. Secondary Outcome: Change From Baseline in Waist Circumference During the Placebo-controlled Period
Time Frame: Baseline and week 2, week 4, and week 16
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Placebo | Apremilast 30 mg
Number analyzed (Participants) | 91 | 185
cm
  Week 2: number analyzed (Participants) | 88 | 174
  Week 2 | -0.2 (3.93) | 0.2 (3.49)
  Week 4: number analyzed (Participants) | 79 | 168
  Week 4 | -0.1 (4.89) | -0.3 (3.63)
  Week 16: number analyzed (Participants) | 67 | 151
  Week 16 | 0.1 (6.16) | -0.9 (5.06)

20. Secondary Outcome: Percentage of Participants Who Achieved a ≥ 4-point Reduction From Baseline in DLQI at Weeks 32 and 52
Description: as for outcome 1
Time Frame: Baseline, week 32 and week 52
Population: Randomized participants who entered the apremilast extension phase. Missing data were imputed using non-responder imputation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo / Apremilast 30 mg: Participants received placebo tablets orally twice a day for 16 weeks followed by 30 mg apremilast orally twice a day from week 16 to week 52.
- Apremilast 30 mg: Participants received 30 mg apremilast tablets orally twice a day for 52 weeks.
Arm/Group | Placebo / Apremilast 30 mg | Apremilast 30 mg
Number analyzed (Participants) | 69 | 152
percentage of participants
  Week 32 | 68.1 [55.8 to 78.8] | 68.4 [60.4 to 75.7]
  Week 52 | 76.8 [65.1 to 86.1] | 79.6 [72.3 to 85.7]

21. Secondary Outcome: Change From Baseline in DLQI at Weeks 32 and 52
Description: as for outcome 2
Time Frame: Baseline, week 32 and week 52
Population: Randomized participants who entered the apremilast extension phase with available data at baseline and each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo / Apremilast 30 mg | Apremilast 30 mg
Number analyzed (Participants) | 69 | 152
score on a scale
  Week 32: number analyzed (Participants) | 62 | 127
  Week 32 | -9.8 (8.19) | -9.9 (7.28)
  Week 52: number analyzed (Participants) | 55 | 112
  Week 52 | -11.3 (7.84) | -11.2 (7.08)

22. Secondary Outcome: Change From Baseline in Itch NRS Score at Weeks 32 and 52
Description: as for outcome 4
Time Frame: Baseline, week 32 and week 52
Population: Randomized participants who entered the apremilast extension phase with available data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo / Apremilast 30 mg | Apremilast 30 mg
Number analyzed (Participants) | 69 | 151
score on a scale
  Week 32: number analyzed (Participants) | 62 | 127
  Week 32 | -3.2 (3.50) | -2.8 (3.22)
  Week 52: number analyzed (Participants) | 54 | 112
  Week 52 | -3.9 (3.61) | -3.3 (3.19)

23. Secondary Outcome: Change From Baseline in Skin Discomfort/Pain VAS at Weeks 32 and 52
Description: as for outcome 5
Time Frame: Baseline, week 32 and week 52
Population: Randomized participants who entered the apremilast extension phase with available data at baseline and each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo / Apremilast 30 mg | Apremilast 30 mg
Number analyzed (Participants) | 69 | 151
score on a scale
  Week 32: number analyzed (Participants) | 57 | 114
  Week 32 | -28.4 (38.40) | -22.6 (33.71)
  Week 52: number analyzed (Participants) | 51 | 104
  Week 52 | -35.0 (36.76) | -31.0 (34.77)

24. Secondary Outcome: Percent Change From Baseline in BSA Affected by Psoriasis at Weeks 32 and 52
Description: as for outcome 3
Time Frame: Baseline, week 32 and week 52
Population: Randomized participants who entered the apremilast extension phase with available data at baseline and each time point
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo / Apremilast 30 mg | Apremilast 30 mg
Number analyzed (Participants) | 69 | 152
percent change
  Week 32: number analyzed (Participants) | 57 | 114
  Week 32 | -49.5 (47.35) | -40.2 (51.79)
  Week 52: number analyzed (Participants) | 51 | 104
  Week 52 | -49.9 (53.25) | -32.0 (93.09)

25. Secondary Outcome: Percentage of Participants Who Achieved a PBI Score of ≥ 1 at Weeks 32 and 52
Description: The PBI is a validated patient-reported instrument to assess patient-relevant benefits of psoriasis treatment. Prior to starting study treatment, participants were asked to assess the importance of a series of treatment goals (from not important to very important) by completing the Patient Needs Questionnaire (PNQ). After a period of treatment (32 weeks and 52 weeks), participants were then asked to assess the extent to which these goals were achieved (from not at all to very) by completing the Patient Benefit Questionnaire (PBQ). The Patient Benefit Index represents the benefits realized as a function of most important needs. The PBI score ranges from 0 (no benefit) to 4 (maximum benefit).
Time Frame: Week 32 and week 52
Population: as for outcome 20
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Apremilast 30 mg | Apremilast 30 mg
Number analyzed (Participants) | 69 | 152
percentage of participants
  Week 32 | 66.7 [54.3 to 77.6] | 67.8 [59.7 to 75.1]
  Week 52 | 65.2 [52.8 to 76.3] | 63.8 [55.6 to 71.4]

26. Secondary Outcome: Percentage of Participants Who Achieved a PASI Score < 3 at Weeks 32 and 52
Description: as for outcome 6
Time Frame: Week 32 and week 52
Population: as for outcome 20
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Apremilast 30 mg | Apremilast 30 mg
Number analyzed (Participants) | 69 | 152
percentage of participants
  Week 32 | 58.0 [45.5 to 69.8] | 40.1 [32.3 to 48.4]
  Week 52 | 50.7 [38.4 to 63.0] | 37.5 [29.8 to 45.7]

27. Secondary Outcome: Percent Change From Baseline in EQ-5D VAS Score at Week 52
Description: as for outcome 8
Time Frame: Baseline and week 52
Population: Randomized participants who entered the apremilast extension phase with available data at baseline and week 52
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo / Apremilast 30 mg | Apremilast 30 mg
Number analyzed (Participants) | 54 | 112
percent change | 51.4 (132.13) | 33.6 (78.53)

28. Secondary Outcome: Percent Change From Baseline in EQ-5D Index Score at Week 52
Description: as for outcome 9
Time Frame: Baseline and week 52
Population: Randomized participants who entered the apremilast extension phase with available data at baseline and week 52
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo / Apremilast 30 mg | Apremilast 30 mg
Number analyzed (Participants) | 54 | 112
percent change | 214.103 (1799.6328) | 11.039 (224.3001)

29. Secondary Outcome: Change From Baseline in WPAI: PSO at Week 52: Percentage Work Time Missed
Description: as for outcome 10
Time Frame: Baseline and week 52
Population: Randomized participants who entered the apremilast extension phase with available data and who had reported being employed at baseline and at week 52.
Measure: Mean (Standard Deviation); unit: percent impairment
Arm/Group | Placebo / Apremilast 30 mg | Apremilast 30 mg
Number analyzed (Participants) | 31 | 64
percent impairment | -4.6 (17.43) | -3.2 (17.11)

30. Secondary Outcome: Change From Baseline in WPAI: PSO at Week 52: Percentage Work Impairment
Description: as for outcome 11
Time Frame: Baseline and week 52
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: percent impairment
Arm/Group | Placebo / Apremilast 30 mg | Apremilast 30 mg
Number analyzed (Participants) | 31 | 64
percent impairment | -21.0 (29.82) | -24.4 (26.78)

31. Secondary Outcome: Change From Baseline in WPAI: PSO at Week 52: Percentage Overall Work Impairment
Description: as for outcome 12
Time Frame: Baseline and week 52
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: percent impairment
Arm/Group | Placebo / Apremilast 30 mg | Apremilast 30 mg
Number analyzed (Participants) | 31 | 64
percent impairment | -21.7 (30.12) | -25.3 (29.91)

32. Secondary Outcome: Change From Baseline in WPAI: PSO at Week 52: Percentage Activity Impairment
Description: as for outcome 13
Time Frame: Baseline and week 52
Population: Randomized participants who entered the apremilast extension phase with available data at baseline and week 52
Measure: Mean (Standard Deviation); unit: percent impairment
Arm/Group | Placebo / Apremilast 30 mg | Apremilast 30 mg
Number analyzed (Participants) | 33 | 75
percent impairment | -32.7 (33.94) | -30.5 (27.01)

33. Secondary Outcome: Number of Participants With TEAEs During Apremilast Treatment
Description: An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values, regardless of etiology. Any worsening of a preexisting condition was considered an AE.
  A serious adverse event (SAE) is any AE occurring at any dose that:
  * Resulted in death;
  * Was life-threatening;
  * Required inpatient hospitalization or prolongation of existing hospitalization;
  * Resulted in persistent or significant disability/incapacity;
  * Was a congenital anomaly/birth defect;
  * Constituted an important medical event. The Investigator assessed the severity/intensity of each event as mild, moderate, or severe based on level of symptoms.
Time Frame: From first dose of apremilast up to 28 days after last dose; up to 40 weeks for participants initially randomized to placebo and 56 weeks for participants initially randomized to apremilast.
Population: All randomized participants who received at least one dose of apremilast, ie, participants originally randomized to apremilast and participants originally randomized to placebo who entered the apremilast extension phase and received at least one dose of apremilast.
Measure: Count of Participants; unit: Participants
Groups:
- Apremilast 30 mg: Participants initially randomized to placebo received apremilast 30 mg orally twice a day from week 16 to week 52. Participants initially randomized to apremilast received apremilast 30 mg orally twice a day for 52 weeks.
Arm/Group | Apremilast 30 mg
Number analyzed (Participants) | 254
Participants
  Any TEAE | 217
  Drug-related TEAE | 152
  Severe TEAEs | 14
  Serious TEAEs | 18
  Serious drug-related TEAE | 2
  TEAE leading to drug interruption | 19
  TEAE leading to drug withdrawal | 31
  TEAE leading to death | 0

34. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities During Apremilast Treatment
Time Frame: as for outcome 33
Population: Randomized participants who received at least 1 dose of apremilast, ie, participants originally randomized to apremilast and participants originally randomized to placebo who entered the apremilast extension phase with at least 1 treatment of apremilast, and with at least 1 post-baseline measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Apremilast 30 mg
Number analyzed (Participants) | 235
Participants
  Alanine Aminotransferase > 3 × ULN | 2
  Albumin < 25 g/L | 0
  Alkaline Phosphatase > 400 U/L | 0
  Aspartate Aminotransferase > 3 × ULN: number analyzed (Participants) | 234
  Aspartate Aminotransferase > 3 × ULN | 1
  Bilirubin > 1.8 × ULN | 1
  Blood Urea Nitrogen > 15 mmol/L | 2
  Calcium < 1.8 mmol/L | 1
  Calcium > 3.0 mmol/L | 0
  Cholesterol > 7.8 mmol/L | 3
  Creatinine > 1.7 × ULN | 1
  Glucose < 2.8 mmol/L | 0
  Glucose > 13.9 mmol/L | 7
  Hemoglobin A1C (Fasting) > 9%: number analyzed (Participants) | 142
  Hemoglobin A1C (Fasting) > 9% | 3
  Lactate Dehydrogenase > 3 × ULN: number analyzed (Participants) | 228
  Lactate Dehydrogenase > 3 × ULN | 0
  Potassium < 3.0 mmol/L | 0
  Potassium > 5.5 mmol/L | 2
  Sodium < 130 mmol/L | 0
  Sodium > 150 mmol/L | 0
  Triglycerides > 3.4 mmol/L | 22
  Hemoglobin: Female < 85 g/L, Male < 105 g/L: number analyzed (Participants) | 232
  Hemoglobin: Female < 85 g/L, Male < 105 g/L | 1
  Hemoglobin: Female > 170 g/L, Male > 185 g/L: number analyzed (Participants) | 232
  Hemoglobin: Female > 170 g/L, Male > 185 g/L | 0
  Leukocytes < 1.5 × 10^9/L: number analyzed (Participants) | 232
  Leukocytes < 1.5 × 10^9/L | 0
  Lymphocytes < 0.8 × 10^9/L: number analyzed (Participants) | 232
  Lymphocytes < 0.8 × 10^9/L | 3
  Neutrophils, Segmented < 1.0 × 10^9/L: number analyzed (Participants) | 232
  Neutrophils, Segmented < 1.0 × 10^9/L | 0
  Platelets < 75 × 10^9/L: number analyzed (Participants) | 232
  Platelets < 75 × 10^9/L | 2
  Platelets > 600 × 10^9/L: number analyzed (Participants) | 232
  Platelets > 600 × 10^9/L | 0

35. Secondary Outcome: Change From Baseline in Blood Pressure at End of Apremilast Extension Period
Time Frame: Baseline (defined as the last value measured on or before the day of the first apremilast dose) and end of apremilast extension period; week 52, or earlier for participants who discontinued prior to week 52
Population: Randomized participants who received at least 1 dose of apremilast, ie, participants originally randomized to apremilast and participants originally randomized to placebo who entered the apremilast extension phase, with a baseline value and at least 1 post-baseline value.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Apremilast 30 mg
Number analyzed (Participants) | 246
mmHg
  Systolic | 0.1 (13.68)
  Diastolic | 0.1 (8.98)

36. Secondary Outcome: Change From Baseline in Pulse Rate at End of Apremilast Extension Period
Time Frame: as for outcome 35
Population: Randomized participants who received at least 1 dose of apremilast, ie, participants originally randomized to apremilast and participants originally randomized to placebo who entered the apremilast extension phase with at least 1 treatment of apremilast, with a baseline value and at least 1 post-baseline value.
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Apremilast 30 mg
Number analyzed (Participants) | 246
beats/minute | 1.0 (10.29)

37. Secondary Outcome: Change From Baseline in Body Weight at End of Apremilast Extension Period
Time Frame: as for outcome 35
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Apremilast 30 mg
Number analyzed (Participants) | 246
kg | -1.20 (3.802)

38. Secondary Outcome: Change From Baseline in Waist Circumference at End of Apremilast Extension Period
Time Frame: as for outcome 35
Population: Baseline and end of apremilast extension period; week 52, or earlier for participants who discontinued prior to week 52
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Apremilast 30 mg
Number analyzed (Participants) | 246
cm | -0.8 (4.97)

ADVERSE EVENTS:
Time Frame: Placebo-controlled period: From first dose of study drug to week 16 or up to 28 days after last dose for participants who didn't enter the apremilast extension period. Apremilast extension period: From first dose of apremilast in the extension period to 28 days after last dose, up to 40 weeks.
Description: All-cause mortality is reported for all participants randomized in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Groups:
- Placebo-controlled Period: Placebo: Participants received placebo tablets orally twice a day for 16 weeks.
- Placebo-controlled Period: Apremilast 30 mg: Participants received apremilast 30 mg tablets orally twice a day for 16 weeks.
- Apremilast Extension Period: Apremilast 30 mg: Participants received apremilast 30 mg tablets orally twice a day from week 16 to week 52 (36 weeks).
Arm/Group | Placebo-controlled Period: Placebo | Placebo-controlled Period: Apremilast 30 mg | Apremilast Extension Period: Apremilast 30 mg
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/185 | 0/221
Serious Adverse Events (participants affected / at risk) | 0/92 | 8/185 | 12/221
Other Adverse Events (participants affected / at risk) | 38/92 | 113/185 | 93/221
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-controlled Period: Placebo (N=92) | Placebo-controlled Period: Apremilast 30 mg (N=185) | Apremilast Extension Period: Apremilast 30 mg (N=221)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Iridocyclitis (Eye disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 2 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 1
Erythema migrans (Infections and infestations) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prolactin-producing pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Varicose vein (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-controlled Period: Placebo (N=92) | Placebo-controlled Period: Apremilast 30 mg (N=185) | Apremilast Extension Period: Apremilast 30 mg (N=221)
Abdominal pain (Gastrointestinal disorders) | 1 | 10 | 4
Abdominal pain upper (Gastrointestinal disorders) | 4 | 12 | 3
Diarrhoea (Gastrointestinal disorders) | 6 | 61 | 22
Nausea (Gastrointestinal disorders) | 5 | 37 | 10
Nasopharyngitis (Infections and infestations) | 11 | 18 | 25
Headache (Nervous system disorders) | 5 | 37 | 19
Psoriasis (Skin and subcutaneous tissue disorders) | 10 | 5 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 6 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT03774875/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT03774875/SAP_001.pdf